CLINICAL TRIAL: NCT06861244
Title: PNOC031: Protocol for Embryonal Tumor With Multilayered Rosettes (ETMR)
Brief Title: Embryonal Tumor With Multilayered Rosettes
Acronym: PNOC031
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pediatric Neuro-Oncology Consortium (Other); Solving Kids' Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240830; NCI-2025-01764 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Embryonal Tumor With Multilayered Rosettes; Embryonal Tumor With Multilayered Rosettes, Nos
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Pyloric Stenosis, Hypertrophic | interventions — Radiotherapy; Standard of Care; Drug Therapy; Temozolomide; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Cohort 1: Gross-total resection, non-metastatic, early radiotherapy (Experimental): Participants will undergo gross total resection of the tumor prior to enrollment into this cohort. Standard dose induction chemotherapy and 6-weeks of early focal radiotherapy, followed by and a second standard dose induction chemotherapy for a total of 12 weeks of chemotherapy; 18 weeks of treatments in all. Participants will be followed for up to 2 years.
  Interventions: Radiation: Radiotherapy (RT); Drug: Chemotherapy Drug, Cancer - Physician's Choice; Procedure: Non-Investigational Surgical Resection; Drug: Temozolomide; Procedure: Tumor Tissue Sample; Procedure: Blood Sample; Procedure: Cerebrospinal Fluid (CSF) Sample
- Cohort 2: Gross-total resection, non-metastatic, high-dose chemotherapy (Experimental): Participants will undergo gross total resection of the tumor prior to enrollment into this cohort. Participants will receive 6 weeks of induction chemotherapy and 3 cycles (approximately 4 weeks each) of high-dose chemotherapy with stem cell rescue and will have the option to receive radiotherapy at the completion of therapy, for a total of 18-24 weeks. Participants will be followed for up to 2 years.
  Interventions: Radiation: Radiotherapy (RT); Drug: Chemotherapy Drug, Cancer - Physician's Choice; Procedure: Non-Investigational Surgical Resection; Drug: Temozolomide; Procedure: Tumor Tissue Sample; Procedure: Blood Sample; Procedure: Cerebrospinal Fluid (CSF) Sample
- Cohort 3A: Metastatic or residual disease, early radiotherapy (Experimental): Participants metastatic disease or residual disease following their initial surgical interventions prior to enrollment into this cohort will receive standard dose induction chemotherapy and 6-weeks of early focal radiotherapy, followed by and a second standard dose induction chemotherapy for a total of 12 weeks of chemotherapy; 18 weeks of treatments in all. Participants will be followed for up to 5 years.
  Interventions: Radiation: Radiotherapy (RT); Drug: Chemotherapy Drug, Cancer - Physician's Choice; Procedure: Non-Investigational Surgical Resection; Drug: Temozolomide; Procedure: Tumor Tissue Sample; Procedure: Blood Sample; Procedure: Cerebrospinal Fluid (CSF) Sample
- Cohort 3B: Metastatic or residual disease, high-dose chemotherapy (Experimental): Participants metastatic disease or residual disease following their initial surgical interventions prior to enrollment into this cohort. Participants will receive 6 weeks of induction chemotherapy and 3 cycles (approximately 4 weeks each) of high-dose chemotherapy with stem cell rescue and will have the option to receive radiotherapy at the completion of therapy, for a total of 18-24 weeks. Participants will be followed for up to 5 years.
  Interventions: Radiation: Radiotherapy (RT); Drug: Chemotherapy Drug, Cancer - Physician's Choice; Procedure: Non-Investigational Surgical Resection; Drug: Temozolomide; Procedure: Tumor Tissue Sample; Procedure: Blood Sample; Procedure: Cerebrospinal Fluid (CSF) Sample

INTERVENTIONS:
Radiation: Radiotherapy (RT) — Undergo RT
  Other Names: Focal Radiotherapy; Radiation Therapy
Drug: Chemotherapy Drug, Cancer - Physician's Choice — One or more of the following may be assigned by the physician (physician's choice) per standard of care guidelines upon study enrollment following surgery: Cytarabine, Carboplatin, Cisplatin, Vincristine Sulfate injection (Vincristine PFS), Topotecan Hydrochloride, Dactinomycin, Thiotepa, Filgrastim, Cyclophosphamide, or Doxorubicin Hydrochloride. Not all participants will receive all possible drug regimens.
  Other Names: Standard of Care, High dose Chemotherapy
Procedure: Non-Investigational Surgical Resection — Undergo surgery directly before study enrollment as part of planned care.
  Other Names: Standard of Care Surgical Resection; Standard of Care Surgical Resection of Tumor
Drug: Temozolomide — Participants assigned to or whom receive optional RT will receive concurrent temozolomide
  Other Names: Temodar
Procedure: Tumor Tissue Sample — Tumor tissue will be collected for correlative studies
  Other Names: Tumor Specimen
Procedure: Blood Sample — Blood samples will be collected for correlative studies
  Other Names: Blood Specimen
Procedure: Cerebrospinal Fluid (CSF) Sample — CSF samples will be collected for correlative studies
  Other Names: CSF Specimen

SUMMARY:
This is an open-label, comprehensive, iterative investigation of evaluating the use of induction chemotherapy, high-dose chemotherapy, and focal radiation therapy in children with newly diagnosed Embryonal Tumor With Multilayered Rosettes (ETMR).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To determine the six-month progression-free survival (PFS6) of participants with newly diagnosed, gross-totally resected, non-metastatic ETMR, treated using a regimen of induction chemotherapy and early focal radiotherapy (Cohort 1)

SECONDARY OBJECTIVES I. To determine the two-year progression-free survival (PFS) and overall survival (OS) of participants with newly diagnosed, gross-totally resected, non-metastatic ETMR (Cohort 1).

II. To determine the two-year progression-free survival (PFS) and overall survival (OS) of participants with newly diagnosed, gross-totally resected, non-metastatic ETMR (Cohort 2).

III. To determine the two-year progression-free survival (PFS), overall survival (OS) and objective response rate of participants with newly diagnosed, incompletely resected and/or metastatic ETMR (Cohort 3A and 3B)

EXPLORATORY OBJECTIVES:

I. To validate the utility of a liquid miRNA biomarker in blood and Cerebral spinal fluid (CSF) as a correlative marker of a participant's disease status.

II. To better define the genomic landscape of ETMR.

OUTLINE:

Participants with newly diagnosed ETMR will obtain either gross total, or sub-total resection surgery prior to enrollment. After surgery, participants will be assigned to 1 of 4 possible cohorts:

Cohorts 1 and 2: Participants with newly diagnosed, gross-totally resected, non-metastatic ETMR.

Cohorts 3A and 3B: Participants with newly diagnosed, incompletely resected and/or metastatic ETMR.

Participants will be assessed for survival outcomes for up to 2 years. Follow-up procedures are to be captured under the PNOC COMP protocol. Participants will be followed under the Pediatric Neuro-Oncology Consortium (PNOC) COMP protocol until death or withdrawal from study.

ELIGIBILITY:
The eligibility criteria listed below are interpreted literally and cannot be waived.

Inclusion Criteria:

1. Participants must have either a molecularly or histologically confirmed embryonal tumor with multilayered rosettes.
2. For enrollment, a confirmation of a minimum of 10-20 unstained formalin-fixed paraffin-embedded (FFPE) slides or 1 block (15-20 mg) with tumor content of 40% or greater is required. Anything less must be discussed and approved by the study chairs prior to enrollment.
3. Prior Therapy:

   1. Cohort 1 participants must not have received any prior tumor-directed therapy other than surgical resection.
   2. Cohort 2 and 3 participants may receive tumor-directed therapy prior to enrollment. These participants must be discussed with study chairs prior to enrollment.
4. Participants must not have received prior radiation for treatment of tumor.
5. Participants of any age are eligible.
6. Participants should begin induction chemotherapy within 28 days of the most recent definitive surgical procedure. Participants beginning therapy beyond 28 days from surgery, will need to discuss with study chairs.
7. Cohort specific eligibility

   1. Cohort 1: Gross-total resection, Eligible for early radiotherapy (please see age criteria below), and no evidence of metastatic disease.
   2. Cohort 2: Gross-total resection, high dose chemotherapy (please see age criteria below), and no evidence of metastatic disease.
   3. Cohort 3A: Metastatic or residual disease, and early radiotherapy.
   4. Cohort 3B: Metastatic or residual disease, and high dose chemotherapy.
   5. Radiotherapy Age Criteria (at the time of planned radiation): >12 months of age for participants with infratentorial tumor OR >15 months of age for participants with supratentorial tumor. For participants being treated on radiotherapy-containing arms, the legal parent/guardian or patient and the physician must be willing to allow the use of radiotherapy for treatment.
8. Performance Score: Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants <=16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
9. Organ Function Requirements:

   1. Peripheral absolute neutrophil count (ANC) > 75,000/mm3
   2. Platelet count > 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 72 hours prior to enrollment).
10. Adequate Renal Function defined as:

    a. Serum creatinine < 1.5 x upper limit normal (ULN) based on age and gender.
11. Adequate Liver Function defined as:

    1. Total bilirubin < 1.5 x upper limit of normal (ULN) for age; in presence of Gilbert's syndrome, total bilirubin < 3 x ULN or direct bilirubin < 1.5 x ULN,
    2. alanine aminotransferase (ALT) < 3 x ULN,
    3. aspartate aminotransferase (AST) < 3 x ULN,
12. Adequate Neurologic Function defined as:

    a. Participants with seizure disorder may be enrolled if well controlled. Participants on enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drugs.
13. As chemotherapeutic agents used in this trial are known to be teratogenic, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
14. Participants must be enrolled on PNOC COMP prior to enrollment on PNOC031 if PNOC COMP is open to accrual at the enrolling institution.
15. A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.

Exclusion Criteria

1. Cohort 1 only: Participants who have received any prior tumor-directed therapy other than surgical intervention
2. Participants who are receiving any other tumor directed investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study.
4. Uncontrolled intercurrent illness.
5. Women of childbearing potential must not be pregnant or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression-free survival at 6 months (PFS6) (Cohort 1) | Up to 6 months
  The median PFS6 is defined as the median number of months for participants in Cohort 1 who have remained progression-free from the date of initial surgical resection until 6 months.

SECONDARY OUTCOMES:
Median Progression-free survival at 2 years progression-free survival (PFS) | Up to 2 years
  The median PFS6 is defined as the median number of months for participants by cohort who have remained progression-free from the date of initial surgical resection until 2 years post-surgery.
Median Overall Survival at 2 years (OS) | Up to 2 years
  The median OS is defined as the median number of months for participants by cohort who are still alive from the date of initial surgical resection until 2 years post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Derek Hanson, MD, Study Chair — Hackensack Meridian Health
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with study collaborators
Supporting Information: Study Protocol, SAP
Time Frame: Until study close out